CLINICAL TRIAL: NCT03447028
Title: A Novel Prognostic Risk Factor for Patients Undergoing Radical Prostatectomy: Triglyseride-Glucose (TyG) Index
Brief Title: Effect of TyG Index on Outcomes of Radical Prostatectomy
Acronym: TyG-PCa
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Ozan HORSANALI, Urologist, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: Recepteutrh
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Syndrome; Prostate Cancer; Insulin Resistance
Keywords: Triglyseride-Glucose index; prostate cancer; radical prostatectomy; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Prostatic Neoplasms; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We investigate the association between Triglyserid-Glucose(TyG) index and prostate cancer in patients undergoing radical prostatectomy.

DETAILED DESCRIPTION:
TyG index is calculated with special formula. Patients undergoing radical prostatectomy are divided two groups according to the cut-off level of 8.55 for TyG index.Groups were compared statistically in terms of oncological outcomes and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical prostatectomy for prostate cancer

Exclusion Criteria:

* taking medicines for established diabetes and dyslipidaemia,
* presence of endocrinological disease,
* history of bariatric surgery,
* missing data and patients with uncontrolled follow-up

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male patients undergoing radical prostatectomy
Study Population: patients undergoing radical prostatectomy for prostate cancer between january 2007 and december 2012.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2012-12-30 (Actual); Study Completion 2012-12-30 (Actual)

PRIMARY OUTCOMES:
Oncological outcomes | 5 years
  Effect of TyG index on oncological outcomes of Prostate cancer

SECONDARY OUTCOMES:
Survival | 5 years
  Death date of patient after radical prostatectomy